CLINICAL TRIAL: NCT02367053
Title: A Randomized, Double-blinded Trial of Single Ascending Doses of ZP4207 Administered s.c. or i.m. to HV and a SD of ZP4207 Administered s.c. to Hypoglycemic T1D to Evaluate the Safety, Tolerability, PKs and PDs of ZP4207 as Compared to an Active Comparator
Brief Title: Single Ascending Doses of ZP4207 Administered in HV and in T1D to Evaluate Safety, Tolerability PKs and PDs of ZP4207 Compared to a Comparator
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZP4207-14013
Record Dates: First submitted 2015-02-03; First posted 2015-02-20 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZP4207 (Experimental): single dose of ZP4207 in ascending doses (s.c. and i.m.)
  Interventions: Drug: ZP4207
- native glucagon (Active Comparator): single fixed dose of glucagon
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: ZP4207
  Arms: ZP4207
Drug: Glucagon
  Arms: native glucagon

SUMMARY:
The trial is a randomized, double-blind First in Human trial to evaluate the safety and tolerability of ZP4207 in healthy volunteers (HV) and in insulin-induced hypoglycemic T1D (type 1 diabetes) subjects as compared to native glucagon. The trial includes two parts.

Part 1 includes dose escalation of ZP4207 in cohorts of 8 subjects. In each cohort, subjects will be randomized 3:1 to receive either a single ascending dose of ZP4207 (6 subjects) or a single fixed dose (SD) of native glucagon (2 subjects). The doses will be administered s.c. in 4-5 cohorts and i.m. in 3 cohorts.

Part 2 includes two sequence groups of 10 hypoglycemic T1D subjects. The subjects will be treated with fixed single doses of ZP4207 and native glucagon s.c. in a sequential cross-over design in a randomized treatment order.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject).
2. Male subjects which are healthy for part 1; for part 2 male subjects with T1D
3. Age between 18 and 50 years, both inclusive.
4. Body weight between 70 and 90 kg, both inclusive.
5. Subjects must be in good health according to age (medical history, physical examination, vital signs, ECG, lab assessments), as judged by the investigator
6. A subject who is surgically sterilized or must be willing to refrain from sexual intercourse during the trial and until one month after completion of the trial or if sexually active, using condom and partner practices contraception during the trial and until one month after completion of the trial.

   For part 2, in addition:
7. Male subjects with T1D for at least one year, as defined by the American Diabetes Association.
8. Having been treated with insulin for T1D for at least 1 year.
9. Stable disease with HbA1c < 8.5 %.
10. Stable insulin treatment during participation in trial and 3 month prior to the screening visit.

Exclusion Criteria:

1. Known or suspected allergy to trial product(s) or related products.
2. Previous participation (randomization) in this trial.
3. Receipt of any investigational drug within 3 months prior to screening.
4. A history or presence of cancer, diabetes (part 1 only), or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, hematological, dermatological, venereal, neurological, psychiatric diseases or other major diseases.
5. Clinically significant illness within 4 weeks before screening, as judged by the investigator
6. Carrier of Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies.
7. Positive result of test for HIV antibodies.
8. Any clinically significant abnormal hematology,biochemistry or urinalysis screening tests, as judged by the Investigator.
9. Clinically significant abnormal ECG at screening as evaluated by Investigator.
10. Donation of blood or plasma in the past month, or in excess of 500 ml within 12 weeks prior to screening.
11. A significant history of alcoholism or drug/chemical abuse, or who has a positive result in the urine drug screen, or who consumes more than 28 units of alcohol per week (one unit of alcohol equals about 250 ml of beer, 1 glass of wine, or 20 ml of spirits).
12. Habitual smoking, i.e., daily smoking or more than 7 cigarettes/week within the last 3 months prior to screening. Subjects have to accept refraining from smoking while at the clinical site.
13. Subjects with mental incapacity or language barriers which preclude adequate understanding or cooperation, who are unwilling to participate in the trial, or who in the opinion of the Investigator should not participate in the trial.
14. Surgery or trauma with significant blood loss within the last 2 months prior to screening.
15. Any condition interfering with trial participation or evaluation or that may be hazardous to the subject.

    For part 2, in addition
16. Severe hypoglycemic events within one year prior to screening, as judged by the investigator.
17. Significant changes in basal insulin within 3 weeks before screening, as judged by the investigator.
18. Clinically relevant diabetic complications (macrovascular disease with symptoms of coronary artery disease or peripheral vascular disease, microvascular disease with symptoms of neuropathy, gastroparesis, retinopathy, nephropathy, or poor blood glucose control with polyuria, polydipsia, or weight loss), as judged by the investigator.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Number of participants with adverse events | 28 days
Safety and Tolerability: Changes or findings from baseline in clinical safety laboratory assessments | 28 days
Safety and Tolerability: Changes or findings from baseline in physical examination | 28 days
Safety and Tolerability: Changes or findings from baseline in vital signs | 28 days
Safety and Tolerability: Changes or findings from baseline in ECG | 28 days
Safety and Tolerability: Findings in local tolerability | 28 days

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area under the curve (AUC) from time-point 0 until 300min | 5 hours
Pharmacokinetics: maximum observed concentration of ZP4207 (Cmax) | 5 hours
Pharmacokinetics: time to maximum observed concentration of ZP4207 (tmax) | 5 hours
Pharmacokinetics: terminal elimination rate constant estimated during the terminal phase of ZP4207 (λz) | 5 hours
Pharmacokinetics: the terminal plasma elimination half-life of ZP4207 (t½), | 5 hours
Pharmacokinetics: apparent volume of distribution of ZP4207 based on plasma concentration values (Vz), estimated during the terminal Phase (f): (Vz/f) | 5 hours
Pharmacokinetics: apparent plasma clearance rate of ZP4207(CL) estimated during the terminal Phase (f) | 5 hours
Pharmacokinetics: mean residence time for plasma ZP4207 (MRT) | 5 hours
Pharmacodynamics (PD): Area under the Plasma glucose curve from time-point 0 until 300 min (AUCgluc 0-300) | 5 hours
Pharmacodynamics: maximum observed concentration (Cmax) | 5 hours
Pharmacodynamics: time to maximum observed concentration (tmax)TPG≥70mg/dL | 5 hours
Pharmacodynamics: Time to plasma glucose equal or above (70 mg/dL) | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jax, MD/PhD, Principal Investigator — Profil GmbH
Locations (1):
- Profil GmbH, Neuss, Germany